CLINICAL TRIAL: NCT03666767
Title: Management and Outcomes of Congenital Anomalies in Low-, Middle- and High-Income Countries: A Multi-Centre, International, Prospective Cohort Study
Brief Title: Management and Outcomes of Congenital Anomalies in Low-, Middle- and High-Income Countries
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Miss Naomi Wright, Miss Naomi Wright, King's College London
Other Study IDs: GPSv7.7/6/2018
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Oesophageal Atresia; Congenital Diaphragmatic Hernia; Intestinal Atresia; Gastroschisis; Exomphalos; Anorectal Malformation; Hirschsprung Disease
MeSH Terms: conditions — Esophageal Atresia; Hernias, Diaphragmatic, Congenital; Intestinal Atresia; Gastroschisis; Hernia, Umbilical; Anorectal Malformations; Hirschsprung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Oesophageal atresia (OA) +/- tracheo-oesophageal fistula (TOF)
  Interventions: Other: Comparisons will be made between LMICs and HICs
- Congenital diaphragmatic hernia (CDH)
  Interventions: Other: Comparisons will be made between LMICs and HICs
- Intestinal atresia (IA)
  Interventions: Other: Comparisons will be made between LMICs and HICs
- Gastroschisis
  Interventions: Other: Comparisons will be made between LMICs and HICs
- Exomphalos
  Interventions: Other: Comparisons will be made between LMICs and HICs
- Anorectal malformation (ARM)
  Interventions: Other: Comparisons will be made between LMICs and HICs
- Hirschsprung's disease
  Interventions: Other: Comparisons will be made between LMICs and HICs

INTERVENTIONS:
Other: Comparisons will be made between LMICs and HICs — Countries will be defined as low, middle or high-income using the World Bank classification.

SUMMARY:
This study is a multi-centre, international, prospective cohort study of congenital anomalies to compare outcomes between LMICs and high-income countries (HICs) globally.

DETAILED DESCRIPTION:
Background: Congenital anomalies have risen to become the 5th leading cause of death in children under 5-years of age globally, yet limited literature exists, particularly from low- and middle-income countries (LMICs) where most of these deaths occur.

Aim: To undertake a multi-centre prospective cohort study of congenital anomalies to compare outcomes between LMICs and high-income countries (HICs) globally.

Methods: The Global PaedSurg Research Collaboration will be established consisting of children's surgical care providers from around the world to participate in the study; collaborators will be co-authors of resulting presentations and publication(s). Data will be collected on patients presenting primarily with seven congenital anomalies (oesophageal atresia, congenital diaphragmatic hernia, intestinal atresia, gastroschisis, exomphalos, anorectal malformation and Hirschsprung's disease) for a minimum of one month between Oct 2018 - April 2019. Anonymous data will be collected on patient demographics, clinical status, interventions and outcome. Data will be captured using the secure, online data collection tool REDCap.

The primary outcome will be all-cause in-hospital mortality and the secondary outcomes will be occurrence of post-operative complications. Chi-squared analysis will be used to compare mortality between LMICs and HICs. Multilevel, multivariate logistic regression analysis will be undertaken to identify patient level and hospital level factors affecting outcomes with adjustment for confounding factors. P<0.05 will be deemed significant. Study approval will be sought from all participating centres. Funding has been granted by the Wellcome Trust.

Outcomes: The study aims to be the first large-scale, geographically comprehensive, multi-centre prospective cohort study of a selection of common congenital anomalies to define current management and outcomes globally. Results will be used to aid advocacy and global health prioritisation and inform future interventional studies aimed at improving outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any neonate, infant or child under the age of 16-years, presenting for the first time, with one of the study conditions can be included in the study.
* Children who have NOT previously received any surgery for their condition.
* Children who have received basic resuscitative and supportive care for their condition at a different healthcare facility and then been transferred to the study centre.
* Patients presenting primarily with one of the study conditions who receive palliative care or no care must be included within the study to reflect true outcomes.

Exclusion Criteria:

* Any neonate, infant or child with one of the study conditions who has previously received surgery (including a stoma) for their condition
* If they have recently received surgery for their condition, were discharged and then represented with a complication of the surgery during the study period they should NOT be included in the study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates, infants and children up to 16-years of age presenting for the first time with one of the seven congenital anomalies in the study to institutions in low-, middle- and high-income countries globally.
  All institutions that provide surgical care for the patients being studied can contribute data. Participating institutions will be recruited through convenience sampling with snowballing.
Sampling Method: Non-Probability Sample
Enrollment: 3850 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
All-cause, in-hospital mortality | Mortality whilst in hospital during primary admission, up to a maximum of 30-days following primary intervention or 30-days following presentation for those who do not receive an intervention and are still in hospital.
  This will include all patients in the study, both those who did not receive an intervention and those that did.
  For patient's hospitalised for over 30-days following primary intervention, a 30-day post-primary intervention mortality rate will be utilised.
  For patients who do not receive a primary intervention (conservative generic ward care only) but remain alive and hospitalised at 30-days following primary admission will have this time point used for recording their mortality status for the primary outcome.

SECONDARY OUTCOMES:
Surgical site-infection | Occurring within 30-days of primary intervention
  This is defined by the Centre for Disease Control as including one or more of the following within 30-days of surgery:
  1) purulent drainage from the superficial or deep (fascia or muscle) incision, but not within the organ/ space component of the surgical site OR 2) at least two of: pain or tenderness; localised swelling; redness; heat; fever; AND the incision is opened deliberately to manage infection, spontaneously dehisces or the clinician diagnoses a SSI (negative culture swab excludes this criterion) OR 3) there is an abscess within the wound (clinically or radiologically detected).
Wound dehiscence | Occurring within 30-days of primary intervention
  All layers of the wound open post-operatively
Need for re-intervention | Occurring within 30-days of primary intervention
  Need for a second unplanned intervention within 30-days of the primary intervention.
Condition specific complications | Occurring within 30-days of primary intervention
  OA: pneumonia, mediastinitis, pneumothorax, chylothorax, haemothorax, anastomotic leak, anastomotic stricture, recurrent TOF, other.
  CDH: air leak, chylothorax, recurrence, adhesional obstruction.
  IA: anastomotic leak/ stenosis, short-gut, missed additional atresia, adhesive bowel obstruction.
  Gastroschisis: ischaemic bowel, abdominal compartment syndrome, necrotising enterocolitis.
  Exomphalos: ruptured sac.
  ARM: electrolyte disturbance, high stoma output (over 20mls/kg/day), stoma prolapse/ retraction/ herniation, peri-stoma skin breakdown (or perianal if primary reconstruction was undertaken without a covering stoma), anal stenosis.
  Hirschsprung's disease: enterocolitis, electrolyte disturbance, high stoma output (over 20mls/kg/day), stoma prolapse/ retraction/ herniation, peri-stoma skin breakdown (or perianal if primary pull-through was undertaken without covering stoma), anal stenosis, post-operative obstruction, anastomotic leak.
Condition specific outcome variables | Occurring within 30-days of primary intervention
  Oesophageal atresia: time to first oral feed (in days) and time to full oral feeds (in days)
Length of hospital stay | Maximum 30-days post-intervention or following presentation for those who do not receive an intervention
  In days, including the first and last day. Time from admission to death in patients who do not survive.
30-day post primary intervention mortality | Death within 30-days of primary intervention or 30-days of presentation in those who do not receive an intervention
Ventilation requirement | Occurring within 30-days of primary intervention or admission for those not receiving an intervention
  Need for any ventilation (excluding during anaesthetic for interventions) and duration of ventilation in days
Time to first enteral feed | Occurring within 30-days of primary intervention or admission for those not receiving an intervention
  In days, including the day of the primary intervention and the day when enteral feeds were started.
Time to full enteral feeds | Occurring within 30-days of primary intervention or admission for those not receiving an intervention
  In days, including the day of the primary intervention and the day when full enteral feeds were achieved.
Parenteral nutrition requirement | Occurring within 30-days of primary intervention or admission for those not receiving an intervention
  Need for any parenteral nutrition and total duration of parenteral nutrition in days for those who receive it.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi J Wright, MBChB BSc MRCS DCH MSc, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the main study results, the full anonymised dataset will be shared with all collaborators and made publicly available. At no time during presentation or publication of the study will individual collaborators, institutions or countries be independently identifiable. For the main study publication, all data within low, middle and high-income countries will be pooled for analysis. Following publication of the main study, collaborators from within a country can undertake a sub-analysis of the data from their country, but only if all collaborators who have contributed data from that country agree. Individual country names will not be identifiable on the dataset made publicly available - each country will be represented by a random number. The publicly available anonymised data will be identifiable by continent allowing for continental sub-analyses to be undertaken.
Supporting Information: Study Protocol
Time Frame: Following publication of the main results.

REFERENCES:
- [Derived] Wright NJ; Global PaedSurg Research Collaboration. Management and outcomes of gastrointestinal congenital anomalies in low, middle and high income countries: protocol for a multicentre, international, prospective cohort study. BMJ Open. 2019 Sep 3;9(8):e030452. doi: 10.1136/bmjopen-2019-030452. PMID 31481373